CLINICAL TRIAL: NCT05091840
Title: Cerebral and Renal Oximetry Study in Preterm Patients Who Require Surfactant Administration
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Principal Investigator, Manuel Sanchez Luna, Chief Neonatology Service, Hospital General Universitario Gregorio Marañon
Other Study IDs: Neuro.Neo.4
Record Dates: First submitted 2021-10-13; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Respiratory Distress Syndrome of Prematurity
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients requiring intubation at birth and subsequent surfactant administration
  Interventions: Other: oximetry monitoring
- patients who receive surfactant by LISA
  Interventions: Other: oximetry monitoring

INTERVENTIONS:
Other: oximetry monitoring — monitoring oximetry in both groups using the INVOS™ system 5100C Oximeter

SUMMARY:
Respiratory distress syndrome of prematurity (RDSP) is an acute respiratory condition that occurs in preterm infants due to pulmonary surfactant deficiency.

Exogenous surfactant administration is a crucial therapeutic measure in the management of RDSP, being the 'less invasive surfactant administration technique' (LISA) the gold standard, according to the latest reviews.

Oximetry based on near-infrared spectroscopy is a non-invasive monitoring modality that provides continuous information on the degree of regional hemoglobin saturation present in the underlying tissue, mainly in the venous compartment. It is thus, a reflection of the balance between oxygen supply and demand of oxygen to the tissues.

We intend to perform a prospective analysis of newborns under 32 weeks of gestational age who require surfactant administration, as we wish to study cerebral and renal perfusion by oximetry in the group of patients who receive surfactant by LISA and in the group of patients who receive surfactant via endotracheal tube (patients intubated at birth for stabilization), since there are few data published in the literature.

Our main hypothesis is that the administration of surfactant by LISA technique does not negatively influence cerebral and renal oximetry.

Our secondary hypothesis is that patients requiring intubation at birth will present greater hemodynamic and respiratory instability in the first 72 hours of life, with a greater decrease in cerebral and renal oximetry with the administration of surfactant, compared to the group that does not require intubation at birth.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants less than 32 weeks gestational age requiring surfactant administration

Exclusion Criteria:

* major congenital malformations
* chromosomopathies

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients less than 32 weeks gestational age born in our center (Hospital General Universitario Gregorio Marañon) who require surfactant administration will be included
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-25 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
to evaluate the impact on cerebral and renal oximetry in preterm infants less than 32 weeks who are administered surfactant | oximetry monitoring first 24 hours after birth

REFERENCES:
- [Background] Bellos I, Fitrou G, Panza R, Pandita A. Comparative efficacy of methods for surfactant administration: a network meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2021 Sep;106(5):474-487. doi: 10.1136/archdischild-2020-319763. Epub 2021 Jan 15. PMID 33452218
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433
- [Background] Abdel-Latif ME, Davis PG, Wheeler KI, De Paoli AG, Dargaville PA. Surfactant therapy via thin catheter in preterm infants with or at risk of respiratory distress syndrome. Cochrane Database Syst Rev. 2021 May 10;5(5):CD011672. doi: 10.1002/14651858.CD011672.pub2. PMID 33970483
- [Background] Scott JP, Hoffman GM. Near-infrared spectroscopy: exposing the dark (venous) side of the circulation. Paediatr Anaesth. 2014 Jan;24(1):74-88. doi: 10.1111/pan.12301. Epub 2013 Nov 23. PMID 24267637
- [Background] Sood BG, McLaughlin K, Cortez J. Near-infrared spectroscopy: applications in neonates. Semin Fetal Neonatal Med. 2015 Jun;20(3):164-72. doi: 10.1016/j.siny.2015.03.008. Epub 2015 Apr 29. PMID 25934116
- [Background] Hanke K, Rausch TK, Paul P, Hellwig I, Kramer C, Stichtenoth G, Herz A, Wieg C, Konig IR, Gopel W, Herting E, Hartel C. The effect of less invasive surfactant administration on cerebral oxygenation in preterm infants. Acta Paediatr. 2020 Feb;109(2):291-299. doi: 10.1111/apa.14939. Epub 2019 Sep 5. PMID 31310677
- [Background] Bertini G, Coviello C, Gozzini E, Bianconi T, Bresci C, Leonardi V, Dani C. Change of Cerebral Oxygenation during Surfactant Treatment in Preterm Infants: "LISA" versus "InSurE" Procedures. Neuropediatrics. 2017 Apr;48(2):98-103. doi: 10.1055/s-0037-1598647. Epub 2017 Feb 28. PMID 28245505
- [Background] Rey-Santano C, Mielgo VE, Gomez-Solaetxe MA, Salomone F, Gastiasoro E, Loureiro B. Cerebral oxygenation associated with INSURE versus LISA procedures in surfactant-deficient newborn piglet RDS model. Pediatr Pulmonol. 2019 May;54(5):644-654. doi: 10.1002/ppul.24277. Epub 2019 Feb 18. PMID 30775857
- [Background] Pellicer A, Greisen G, Benders M, Claris O, Dempsey E, Fumagalli M, Gluud C, Hagmann C, Hellstrom-Westas L, Hyttel-Sorensen S, Lemmers P, Naulaers G, Pichler G, Roll C, van Bel F, van Oeveren W, Skoog M, Wolf M, Austin T. The SafeBoosC phase II randomised clinical trial: a treatment guideline for targeted near-infrared-derived cerebral tissue oxygenation versus standard treatment in extremely preterm infants. Neonatology. 2013;104(3):171-8. doi: 10.1159/000351346. Epub 2013 Aug 1. PMID 23921600